CLINICAL TRIAL: NCT07078396
Title: Duration and Analgesic Quality of 1% Ropivacaine Ankle Blocks for Forefoot Surgeries - A Retrospective Analysis
Brief Title: Duration and Quality of 1% Ropivacaine Ankle Blocks
Acronym: AQAB
Status: Completed | Type: Observational
Sponsor: Ziekenhuis Oost-Limburg (Other)
Responsible Party: Principal Investigator, Imré Van Herreweghe, Anesthesiologist, Principle Investigator, Ziekenhuis Oost-Limburg
Other Study IDs: AQAB
Record Dates: First submitted 2025-06-26; First posted 2025-07-22 (Actual); Last update posted 2025-07-22 (Actual); Status verified 2025-07

CONDITIONS: Forefoot Surgery
Keywords: Ultrasound-guided; Ankle block; Ropivacaine; Forefoot surgery; Block duration

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this observational study is to determine the analgesic duration and analgesic quality of a 1% ropivacaine ankle block in forefoot surgery. Bilateral cases of forefoot surgery, preoperative use of steroids, preexisting lower extremity neuropathy, or failed blocks were not included in this quality improvement program.

An ankle block with 1% ropivcaine and patient follow-up is part of the standard practice at Ziekenhuis Oost-Limburg.

ELIGIBILITY:
Inclusion Criteria:

* Patients who underwent unilateral elective forefoot surgery under ankle block with 1% ropivacaine between December 2023 and April 2024 at Ziekenhuis Oost-Limburg, Genk, Belgium.

Exclusion Criteria:

* Bilateral cases of forefoot surgery
* Preoperative use of steroids,
* Preexisting lower extremity neuropathy
* Failed blocks

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Ziekenhuis Oost-Limburg, Genk, Belgium.
Sampling Method: Non-Probability Sample
Enrollment: 56 (Actual)
Dates: Start 2023-12-01 (Actual); Primary Completion 2024-04-24 (Actual); Study Completion 2024-04-30 (Actual)

PRIMARY OUTCOMES:
Duration sensory block | A maximum of 72 hours until return of sensation is expected.
  Every patient was contacted by phone to assess the duration of analgesia, maximum pain scores within the first 24 hours and patient satisfaction with analgesia on a 10-point visual analog scale (VAS), opioid consumption in the first 24 hours, sleep quality, side effects, and ease of mobilization. If the sensory block had not disappeared at the moment of the survey or if the patient could not be reached, the patient was called again the day after.

CONTACTS AND LOCATIONS:
Locations (1):
- Ziekenhuis Oost-Limburg, Genk, Belgium

IPD SHARING:
Plan to Share IPD: No